CLINICAL TRIAL: NCT04999566
Title: Cardiac Manifestations in Adult Patients With Inherited Metabolic Disease: a Case Series
Brief Title: Cardiac Manifestation and Inherited Metabolic Diseases
Status: Completed | Type: Observational
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Christel Tran, Principal Investigator, University of Lausanne
Other Study IDs: 2020-02531
Record Dates: First submitted 2021-07-19; First posted 2021-08-11 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2023-11

CONDITIONS: Metabolism, Inborn Errors
Keywords: Cardiac involvement; Inborn errors of metabolism
MeSH Terms: conditions — Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to report and describe cardiac manifestations associated with IMD in a cohort of patients followed in a reference center for rare diseases (Lausanne University Hospital, CHUV) from 2017-2020.

DETAILED DESCRIPTION:
Inherited metabolic diseases (IMD) are genetic disorders resulting from an enzyme defect and/or transport proteins in metabolic pathways affecting proteins, fat, carbohydrate metabolism or impaired organelle function. As IMDs can affect the primary sources of energy (glycogen, fatty acids), they can lead to cardiac dysfunction. Although most of IMDs are multisystemic diseases, in some cases, the cardiac dysfunction they cause is the main clinical feature and source of major complications which will determine the prognosis, like heart failure, ventricular arrythmias or even sudden death. Information regarding cardiac manifestations in adult IMDs is currently scarce and little is known about their clinical and radiological characteristics.

A database was created in 2017 including all patients with IMD followed at the Adult Metabolic Clinic in the CHUV. This database was part of a protocol submitted and approved by the Ethics committee (# 2017-02328). The results of this first analysis were published in the Journal of Orphan Rare Diseases. Investigators will use this database to identify all the patients who had cardiac examination. Only patients from the Lausanne University Hospital followed jointly with the Division of Cardiology will be included in the analysis. Electronic and paper patient charts from the Division of Genetic Medicine and Division of Cardiology (Lausanne University Hospital) will be reviewed for type of IMD and cardiac investigations (cardiac ultrasound, multiple resonance Imaging, electrocardiogram). All variables will be entered in an excel database.

ELIGIBILITY:
Inclusion Criteria:

* All IMD adult patients followed at the adult metabolic clinic at the Lausanne University Hospital from 2017 to 2020 with cardiac investigations

Exclusion Criteria:

* Age < 16 years. Any document attesting a refusal to participate will exclude the data entry of the concerned patient

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient clinic for Adult patients with inherited metabolic diseases (IMD) from the Lausanne University Hospital (Division of Genetic Medicine)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Specific diagnosis of Inborn Errors of Metabolism listed by their frequency | Day 1
  Clinical outcome
Age at diagnosis (years/months) | Day 1
  Clinical outcome
Current age (years/months) | through study completion, an average of 1 year
  Clinical outcome
Weight (kg) | through study completion, an average of 1 year
  Clinical outcome
Height (cm) | through study completion, an average of 1 year
  Clinical outcome
BMI (kg/m^2) | through study completion, an average of 1 year
  Clinical outcome. Weight and height will be combined to report BMI
Cardiac involvement | 3 years
  Type of complications (restrictive cardiomyopathy, hypertrophic cardiomyopathy, dilated cardiomyopathy, arrythmia, heart failure, valvlulopathy, cardiomegaly, thrombosis)
Left ventricular mass (g/m^2) | 3 years
  Cardiac ultrasound and multiple resonance imaging description of left ventricular mass
Left ventricular volume (cc/m^2) | 3 years
  Cardiac ultrasound and multiple resonance imaging description of left ventricular volume
Right ventricular volume (cc/m^2) | 3 years
  Cardiac ultrasound and multiple resonance imaging description of right ventricular volume
Left ventricular diameter (mm) | 3 years
  Cardiac ultrasound and multiple resonance imaging description of left ventricular diameter
Left ventricular ejection fraction (%) | 3 years
  Cardiac ultrasound and multiple resonance imaging description of left ventricular ejection fraction
Right ventricular ejection fraction (%) | 3 years
  Cardiac ultrasound and multiple resonance imaging description of right ventricular ejection fraction
aortic root diameter (mm) | 3 years
  Cardiac ultrasound and multiple resonance imaging description of aortic root diameter
Additional cardiac investigations | 3 years
  ECG-QT interval

SECONDARY OUTCOMES:
Specific treatment for inherited metabolic diseases | 3 years
  Treatment specific to each diseases including ammonia scavenger, enzyme replacement therapy, vitamin cofactors
Gender (Male/Female) | Day 1
  Demography outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Gariani K, Nascimento M, Superti-Furga A, Tran C. Clouds over IMD? Perspectives for inherited metabolic diseases in adults from a retrospective cohort study in two Swiss adult metabolic clinics. Orphanet J Rare Dis. 2020 Aug 18;15(1):210. doi: 10.1186/s13023-020-01471-z. PMID 32811506
- See also: Article open-access — https://pubmed.ncbi.nlm.nih.gov/32811506/